CLINICAL TRIAL: NCT07338474
Title: Postoperative Physical Activity and Posture in Patients Undergoing Enhanced Recovery Video-Assisted Thoracoscopic Lobectomy and Segmentectomy
Brief Title: Mobilization Before and After Video-Assisted Thoracoscopic Surgery Lobectomy/Segmentectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lasse Visby, Medical Doctor, Rigshospitalet, Denmark
Other Study IDs: P-2024-17015
Record Dates: First submitted 2025-10-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (NSCLC); Perioperative Care; Enhanced Recovery After Surgery
Keywords: mobilization; ERAS; posture; minimizing complications; fast-track; lung-surgery; thoracic-surgery
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine mobilization before/after Video-Assisted Thoracoscopic Surgery Lobectomy/Segmentectomy and further assess possible barriers to mobilization.

DETAILED DESCRIPTION:
50 patients will be included in the study. Patients will wear a SENS motion, accelerometer for minimum 48 hours before surgery and until discharge (or maximum 7 days). Mobilization and posture will be measured 24h. Twice daily the patients will be assessed with a multidimensional questionnaire about barriers to mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to understand written and spoken Danish language
* Signed written informed consent form.
* Patient planned to elective VATS lobectomy or segmentectomy
* Patients with the pre-operative examination done minimum 48 hours prior to surgery (to allow at least 48 hours of preoperative activity monitoring)

Exclusion Criteria:

* Patients with diagnoses (neurological, psychiatric, orthopedic etc.) that challenges postoperative mobilization and posture changes.
* Patient undergoing re-surgery
* Patients admitted to intensive care unit
* Patients with a conversion to open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing VATS lobectomy/segmentectomy at the Department of Cardiothoracic Surgery, Rigshospitalet, Denmark, that adheres to the above inclusion/exclusion criterias
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-05-03 (Actual)

PRIMARY OUTCOMES:
Minutes spent supine, sitting and standing | Before surgery: From enrollment to surgery day (minimum 48 hours) and After surgery: From 3 hours post surgery and until discharge or maximum 7 days.

SECONDARY OUTCOMES:
Time spent out of bed | Before surgery: From enrollment to surgery day (minimum 48 hours) and After surgery: From 3 hours post surgery and until discharge or maximum 7 days.
Pulmonary complications | Within 30 days
Length of hospital stay | Days counted after surgery. Day of surgery is day 0.
Reasons for not being mobilized (questionnaire) | Filled out twice daily on first and second postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No